CLINICAL TRIAL: NCT03622008
Title: A Phase 1, Randomized, Double-Blind Study to Investigate the Multiple Dose Safety, Tolerability and Pharmacokinetics of WCK 4282 (FEP-TAZ) After Intravenous Administrations in Healthy Volunteers
Brief Title: To Investigate the Multiple Dose Safety, Tolerability and Pharmacokinetics of WCK 4282 (FEP-TAZ)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Clinartis, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: W-4282-105
Record Dates: First submitted 2018-07-15; First posted 2018-08-09 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Antibiotics Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Intervention Model Description: Subjects will receive one of the following IV treatments as a q8h infusion (90 min) regimen for 10 days:
  * FEP-TAZ 4 g (2 g cefepime + 2 g tazobactam) (n=16)
  * Placebo (n=4)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FEP-TAZ 4 g (Experimental): FEP-TAZ 4 g (2 g cefepime + 2 g tazobactam) IV treatments as a q8h infusion (90 min) regimen for 10 days
  Interventions: Drug: FEP-TAZ 4 g
- Placebo (Placebo Comparator): placebo IV
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FEP-TAZ 4 g — FEP-TAZ 4 g (2 g cefepime + 2 g tazobactam) IV treatments as a q8h infusion (90 min) regimen for 10 days
  Arms: FEP-TAZ 4 g
Other: Placebo — Placebo IV
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetics (PK) of multiple IV doses of FEP-TAZ 4 g (2 g cefepime + 2 g tazobactam) administered every 8 hours (q8h) in healthy adult volunteers for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a body Mass Index (BMI) between 18 to 32 kg/m2 (both inclusive).
* Medical history without any major pathology.
* A sustained supine systolic blood pressure <150 mm Hg or >90 mm Hg or a supine diastolic blood pressure <95 mm Hg or >50 mm Hg at Screening or Check-in (Day -1). Blood pressure may be retested once in the supine position.
* Glomerular filtration rate (GFR) > 80 mL/min, estimated by the Cockcroft-Gault equation.

Exclusion Criteria:

* Use of cefepime and/or tazobactam within 60 days prior to study drug administration.
* History or evidence of clinically relevant pathology which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-05-13 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Safety assessed by number of abnormal clinical laboratory test result | every 8 hours
To measure the Maximum Concentration | 24 hrs
To measure the Area Under the Curve [AUC] | 24 hrs
Safety assessed by number of abnormal physical examinations findings. | every 8 hours
Safety assessed by number of abnormal vital signs findings | every 8 hours
Safety assessed by number of abnormal 12 Lead ECG findings | every 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States